CLINICAL TRIAL: NCT01914055
Title: Dissecting the Role of Distal Embolization of Athero-thrombotic Material in Primary PCI: the ThrombOticBurden and mIcrovAscularobStruction (TOBIAS) Study.
Acronym: TOBIAS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale San Donato (Other)
Responsible Party: Principal Investigator, Leonardo Bolognese, MD, Director, Ospedale San Donato
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Arezzo009
Record Dates: First submitted 2013-07-12; First posted 2013-08-01 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- angio-guided thrombus aspiration (Active Comparator): thrombus aspiration guided by angiography
  Interventions: Device: angio-guided thrombus aspiration (Eliminate catheter, Terumo, Tokyo, Japan)
- OCT-guided thrombus aspiration (Experimental): thrombus aspiration guided by optical coherence tomography
  Interventions: Device: OCT-guided thrombus aspiration (Eliminate catheter, Terumo, Tokyo, Japan)

INTERVENTIONS:
Device: angio-guided thrombus aspiration (Eliminate catheter, Terumo, Tokyo, Japan) — angio-guided thrombus aspiration with monorail thrombus aspiration catheter (Eliminate, Terumo, Tokyo, Japan)
  Arms: angio-guided thrombus aspiration
Device: OCT-guided thrombus aspiration (Eliminate catheter, Terumo, Tokyo, Japan) — FD-OCT-guided thrombus aspiration with monorail thrombus aspiration catheter (Eliminate, Terumo, Tokyo, Japan); OCT images will be acquired at the site of culprit coronary artery with a commercially available system (Lunawave System; Fastview catheter/Terumo, Tokio, Japan OR C7 System; LightLab Imaging Inc; C7 Dragonfly catheter/St Jude Medical, Westford, MA)
  Arms: OCT-guided thrombus aspiration

SUMMARY:
demonstrate that FD-OCT guidance is feasible and possibly results in reduction of frequency-domain Optical Coherence Tomography-defined residual thrombus burden after thrombus-aspiration.

ELIGIBILITY:
Inclusion Criteria:

* ST elevation myocardial infarction
* Ages Eligible for Study: >18 years old
* Genders Eligible for Study: Both (female sex with child-bearing potential excluded)

Exclusion Criteria:

* occluded (TIMI 0) or sub occluded (TIMI 1) proximal vessel of estimated diameter ≥3mm
* intended use of thrombus aspiration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
number of cross-sections with thrombus area more than 10% at post-stenting frequency-domain (FD) Optical Coherence Tomography | within the primary PCI procedure
  Whether FD-OCT guidance of manual thrombus aspiration (TA) is superior to conventional angio-guided TA in reducing residual thrombus burden after stenting (defined as the number of cross-sections with thrombus area more than 10% at post-stenting FD-OCT)

SECONDARY OUTCOMES:
major adverse cardiac events | at 6 months
  rate of major adverse cardiac events at 6 months from the index procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Department, Ospedale S.Donato, Arezzo, AR, Italy